CLINICAL TRIAL: NCT03270462
Title: A Pilot Study of Stable Kidney Transplant Recipients Taking Tacrolimus With CNS Symptoms Switched to Envarsus
Brief Title: CNS Study of Patients Switching From Tacrolimus to Envarsus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0781
Record Dates: First submitted 2017-08-16; First posted 2017-09-01 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Renal Transplant Patients
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Envarsus XR (Other): A form of the anti-rejection drug, tacrolimus, for people who have had a kidney transplant.
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Envarsus XR — Pilot study documenting the neurotoxic side effects including tremors in patients with stable graft who are receiving Tacrolimus (Envarsus XR) following kidney transplantation. Standardized questionnaire will be used to document these symptoms.
  Other Names: Tacrolimus

SUMMARY:
This is a pilot study documenting the neurotoxic side effects including tremors in patients with a stable graft who are receiving Tacrolimus following kidney transplantation. A standardized questionnaire will be used to document these symptoms.

DETAILED DESCRIPTION:
Immunosuppressive therapies have burdensome side effects which may lead to sub-therapeutic dosing and non-compliance.

This study provides renal transplant patients the opportunity for an alternative treatment using tacrolimus, with possible less Central Nervous Symptom (CNS) side effects. CNS side effects are one of the main reasons that patients complain about after having a kidney transplant while on tacrolimus (Prograf). The side effects can be debilitating and can affect the patient's overall well-being. In severe cases it may lead to non-compliance. The advantage of the study of using Envarsus is the ability to avoid these debilitating CNS side effects and afford better compliance with the patients taking the medicine.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients with stable graft function.
* More than 1 months post-transplant.
* 18+ years of age with some CNS problems secondary to Prograf (tacrolimus).

Exclusion Criteria:

* Multi-organ patients (kidney/pancreas, kidney/liver).
* Evidence of graft rejection or treatment of acute rejection within 14 days prior to baseline visit.
* Inability to self-administer the QOL questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-05-02 (Actual); Study Completion 2020-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Chan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Lisa Kornfeld, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Envarsus XR
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Envarsus XR
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: The Investigators will evaluate the quality of life between baseline and 6 months related to sleep disturbance and upper extremity fine motor skills/ADL (activities of daily living), with the goal to be an improvement in their quality of life. This was assessed via a study-specific clinical assessment that evaluated patient reports of hand tremor and related complaints, and scored in a range of 0 to 3, with higher scores indicating worse symptoms of hand tremor, and a lower QOL.
Time Frame: Baseline, 1 Month, 6 Months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Envarsus XR
Number analyzed (Participants) | 20
score on a scale
  Baseline | 2.7 [2 to 3]
  Month 1 | 1.35 [0 to 2]
  Month 6 | 0.2 [0 to 1]

2. Secondary Outcome: Therapeutic Tacrolimus Drug Levels
Description: The Investigators will evaluate Tacrolimus drug levels and will document any adverse events associated with this measure.
Time Frame: Baseline, 1 Month, 6 Months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Envarsus XR
Number analyzed (Participants) | 20
ng/ml
  Baseline | 8.66 (2.71)
  Month 1 | 8.58 (1.75)
  Month 6 | 8.48 (2.43)

3. Secondary Outcome: Kidney Function: Serum Creatinine Levels
Description: The Investigators will evaluate serum creatinine levels and will document any adverse events associated with this measure.
Time Frame: Baseline, 1 Month, 6 Months
Measure: Geometric Mean (Standard Deviation); unit: mg/dl
Arm/Group | Envarsus XR
Number analyzed (Participants) | 20
mg/dl
  Baseline | 1.19 (0.31)
  Month 1 | 1.14 (0.34)
  Month 6 | 1.11 (0.35)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Envarsus XR
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03270462/Prot_SAP_000.pdf